CLINICAL TRIAL: NCT02543749
Title: Dendritic Cells as Autologous Vaccine in Patients With Chronic Myeloid Leukemia
Brief Title: DC Vaccination in CML
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jörg Westermann, MD, Representative of the sponsor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571ADE60; 2006-006962-41 (EudraCT Number)
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: CML; DC vaccine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC vaccine (Experimental): Autologous DC pulsed with leukemia-associated peptides+adjuvant.
  Ten vaccinations over 26 weeks with 10 x 106 freshly thawed DC Intradermal injections (1-2 ml volume)
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — Autologous DC pulsed with leukemia-associated peptides+adjuvant

SUMMARY:
The aim of this phase I/II trial is induction of anti leukemic T cell immunity in a clinical situation of "minimal residual disease". This might be a strategy to immunologically eradicate the residual leukemia cells. Patients to be included are chronic phase bcr/abl+ CML (chronic myeloid leukemia) patients in stable cytogenetic and/or molecular remission.

These patients can be included if they have:

1. not achieved a CMR (complete molecular response) or
2. achieved bcr/abl < 10% on qPCR (quantitative polymerase chain reaction) (=MCyR) (Major cytogenic Response), but less than a CCyR (complete cytogenic Response).

Autologous DC (Dendritic cells), generated under GMP (Good manufacturing conditions) conditions, are used as a vaccine. These DC constitutively express all putative tumor antigens. In order to ensure sufficient presentation of distinct CML-related antigens, particularly in good responders to TKIs, DC are additionally pulsed with peptides from bcr/abl, WT-1 (Wilms Tumor Protein) and proteinase-3. Monitoring of T cell reactivity against these peptides can then serve as surrogate marker for anti leukemic immunity induced by the vaccine. Vaccination is performed with 10^7 DC i.d. (intra dermal) in weeks 1, 3, 5, 8, 11, 14, 17, 20, 23 and 26. KLH (keyhole limpet hemocyanin) is used as an adjuvant for vaccine preparations in weeks 3, 5 and 8 (and 11).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bcr/abl-positive CML in stable cytogenetic / molecular remission after at least 18 months therapy with tyrosine kinase Inhibitors (TKI). The following groups of patients will be included:

   * complete cytogenetic remission (CCyR), but stable detection of bcr/abl-transcript on qPCR (at least on two different time points over a period of at least 6 months). A stable molecular remission is assumed, if the difference between the qPCR values does not exceed a factor 5 (< 0,5log).
   * No CCyR, but qPCR for bcr/abl transcript < 10% (= MCyR (Major cytogenetic Response)) after at least 24 months on 2nd generation TKI therapy.
2. Treatment with a TKI inhibitor and an additional anti leukemic drug is no exclusion criterion.
3. Age 18-80 years
4. Performance status of 0 or 1 according to WHO index or Karnofsky index >70 %
5. Life expectancy > 18 months
6. Hematological function should be at least partially conserved (platelets count >50.000/ μl, Hb > 8g/dl)
7. written informed consent
8. No breast feeding
9. if of childbearing potential, negative pregnancy test (serum/urine ß- HCG ( human chorionic gonadotropin )) and willingness to use highly effective contraceptive methods (Pearl Index <1, e.g.: birth control pill, loop, hormone implant, transdermal hormone patch, a combination of two barrier methods [condom and vaginal diaphragm] sterilisation or sexual abstinence) for the study duration and thereafter as long as under treatment with antileukemic drugs

Exclusion Criteria:

1. Clinically relevant autoimmune disorders
2. Immunodeficiency syndromes
3. Known allergy to GM-CSF (granulocyte macrophage colony-stimulating factor), TNF-α (Tumor necrosis factor Alpha) , IL-4 (interleukine 4) or KLH (keyhole limpet hemocyanin)
4. Pregnancy (absence confirmed by serum/urine ß-HCG) or breastfeeding
5. Women of childbearing age without highly effective contraception
6. Active infectious disease requiring treatment
7. Continuous therapy with corticosteroids or other immunosuppressive drugs
8. Severe psychiatric disorders
9. Organ dysfunction:

   * Thrombin Time / Partial Thromboplastin Time > 1,5 x upper normal limit
   * creatinine > 2,0 mg/ml
   * Bilirubin > 3,0 mg/ml, ALAT/ASAT (Alanine aminotransferase/ aspartate aminotransferase) > 3x upper normal limit
   * pulmonary disfunction (dyspnea at rest or with minimal exertion)
   * clinically relevant coronary heart disease or ventricular arrhythmia, congestive heart failure > grade II NYHA (New York Heart Association)
10. Persons who are detained officially or legally to an official institute
11. Subjects for whom there is concern about compliance with the protocol procedures
12. Present History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) that could limit the subject's ability to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
DC toxicity Parameters using CTC (Common toxicity criteria) | 30 weeks
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 (Treatment: long-term vaccination with peptide-pulsed autologous DC in patients with chronic phase CML who have persistent residual cytogenetic and/or molecular disease after at least 18 months therapy with a tyrosine kinase Inhibitor)

SECONDARY OUTCOMES:
Molecular/cytogenetic Response under vaccination as measured by qPCR for bcr/abl in % IS (International scale) | 30 weeks
T-cell Response: Antigen specific T-cell Response in % CD8+ T-cells for bcr/abl | 30 weeks
T-cell Response: Antigen specific T-cell Response in % CD4+ T-cells for bcr/abl | 30 weeks
T-cell Response: Antigen specific T-cell Response in % CD8+ T-cells for WT-1 (only in HLA-A2+ patients) | 30 weeks
T-cell Response: Antigen specific T-cell Response in % CD8+ T-cells for Proteinase 3 (only in HLA-A2+ patients) | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J. Westermann, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité - University Medicine Berlin, Berlin
  - Klinikum Bremen Mitte, Bremen